CLINICAL TRIAL: NCT07117396
Title: Clinical and Laboratory Predictors of Chronic Pain After Critical Illness: A Prospective Analysis of Intensive Care Unit Survivors
Brief Title: Chronic Pain After Intensive Care Unit: Clinical Predictors
Status: Completed | Type: Observational
Sponsor: Attikon Hospital (Other)
Responsible Party: Principal Investigator, Milionis Orestis, Principal Investigator, Attikon Hospital
Other Study IDs: AttikonH 09.10.2024
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: ICU Hospitalization; Chronic Pain
Keywords: ICU Hospitalization; Chronic pain; Predictors
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Thanks to medical advances, more patients now survive their stay in the Intensive Care Unit (ICU). However, many people who leave the ICU face long-term health problems, known as Post-Intensive Care Syndrome (PICS). This can include physical weakness, memory or thinking problems, anxiety or depression - and chronic pain.

Chronic pain is pain that lasts more than 12 weeks and can interfere with your daily life. Studies show that many ICU survivors still experience moderate to severe pain even a year after they go home, especially in the shoulders. This pain is often linked to conditions like severe infections or older age, but it's not yet fully understood.

To help improve care, researchers at Attikon University Hospital in Athens are studying ICU survivors to learn:

How common chronic pain is

Where it appears in the body

How severe it is

How it affects everyday activities

They are also looking at health history, treatments received in the ICU, and lab results to see if any of these are linked to pain after discharge.

If you or your loved one has been in the ICU and experiences ongoing pain, know that you're not alone - and that researchers and doctors are working to better understand and manage this problem.

DETAILED DESCRIPTION:
Over the past two decades, improved intensive care practices have significantly reduced in-hospital mortality. However, a growing number of survivors experience a range of long-term complications, collectively known as Post-Intensive Care Syndrome (PICS). A key but underexplored component of PICS is chronic pain, defined as persistent pain lasting beyond 12 weeks or beyond the expected healing time following trauma or surgery.

Existing data suggest that up to 73% of ICU survivors report moderate to severe pain one year after discharge, with the shoulder being the most commonly affected anatomical region. Retrospective studies estimate the prevalence of chronic pain among ICU survivors to be as high as 44%. Identified risk factors include advanced age and severe sepsis; however, there is limited evidence regarding the true impact of chronic pain on activities of daily living (ADLs), its intensity, and clinical predictors.

This prospective observational study is conducted at the Intensive Care Unit of Attikon General University Hospital in Athens, Greece, and includes both medical and surgical ICU patients, including cardiothoracic surgery cases. The aim is to assess the prevalence, anatomical distribution, and intensity of chronic pain in ICU survivors, examine its interference with daily functioning, and explore associations between chronic pain and clinical or laboratory data collected during ICU admission, hospitalization, and discharge.

Patients are evaluated at three timepoints: ICU admission, ICU discharge, and three months post-ICU discharge. The inclusion criteria are age ≥18 years and ICU stay of at least 24 hours.

Detailed data collection includes:

Demographics and Lifestyle: Age, sex, educational level, occupation, weight, height, Body Mass Index (BMI), weekly physical activity.

Pain History and Characteristics: Prior history of chronic or acute pain, anatomical localization, intensity with Visual Analogue Scale score (VAS score), and pain qualities assessed using the validated Greek version of the Short-Form McGill Pain Questionnaire.

Medical History: Hypertension, dyslipidemia, arrhythmias, coronary artery disease, Chronic Obstructive Pulmonary Disease (COPD), Asthma, Obstructive Sleep Apnoea (OSA), chronic kidney disease, Gastro Esophageal Reflux Disease (GERD), peptic ulcer, thyroid disorders, diabetes, stroke, migraine, epilepsy, musculoskeletal/rheumatologic conditions, psychiatric disorders, surgical history, and opioid use.

ICU Parameters: Duration of stay, use of vasopressors, sedatives, opioids, presence of sepsis, mechanical ventilation,Acure Respiratory Distress Syndrome (ARDS), surgical procedures, and regional anesthesia.

Laboratory Data at ICU Admission and Discharge: Hematocrit, hemoglobin, White Blood Cell count (WBC), platelets, International Normalized Ratio (INR), C-reactive protein (CRP) ,fibrinogen, procalcitonin, creatinine, urea, potential of hydrogen (pH), Partial pressure of carbon dioxide (pCO₂), Partial pressure of oxygen (pO₂), Bicarbonate (HCO₃-), potassium, sodium, calcium, phosphorus, magnesium, chloride, Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), Gamma-Glutamyl Transferase (GGT), Alkaline Phosphatase (ALP), total bilirubin, albumin, and Thyroid-Stimulating Hormone (TSH).

The study's overarching goal is to better characterize the burden of chronic pain among ICU survivors and to inform the development of targeted preventive and therapeutic strategies. Ethical approval has been granted by the Institutional Ethics Committee of Attikon University Hospital, and all participants provide written informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years old and
* A minimum of one day of intensive care unit (ICU) hospitalization

Exclusion Criteria:

* Age less than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Both medical and surgical patients. All eligible individuals assessed at three distinct timepoints: upon ICU admission, at ICU discharge, and three months following ICU discharge.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2024-10-11 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Chronic pain | three months post discharge
  Assement of chronic pain via questionnaire (Short-form McGill Pain Questionnaire)

CONTACTS AND LOCATIONS:
Locations (1):
- Attikon University Hospital, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: Undecided